CLINICAL TRIAL: NCT04631965
Title: Bridge: an International Longitudinal Study of Healthcare Transition of Adolescents With Severe Chronic Health Conditions
Brief Title: Healthcare Transition of Adolescents With Chronic Health Conditions
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Collaborators: Pediatric Research Center (Unknown); Foundation for Medical Research (Other); Foundation for Paediatric Research, Finland (Other); The Paulo Foundation (Other); Royal Children's Hospital (Other); Murdoch Childrens Research Institute (Other); University of Melbourne (Other)
Responsible Party: Principal Investigator, Silja Kosola, MD PhD, Adjunct professor in Adolescent Medicine, University of Helsinki
Other Study IDs: U1011SILTA
Record Dates: First submitted 2020-10-21; First posted 2020-11-17 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Transition; Diabetes; Kidney Diseases; Liver Diseases; Inflammatory Bowel Diseases; Rheumatic Diseases; Congenital Heart Disease; Neurologic Disorder
Keywords: adolescent
MeSH Terms: conditions — Diabetes Mellitus; Kidney Diseases; Liver Diseases; Inflammatory Bowel Diseases; Rheumatic Diseases; Heart Defects, Congenital; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort in Finland: 253 young patients who attend clinics in Finland with no hospital-wide transition support service available
- Cohort in Australia: 250 young patients who attend clinics in Victoria, Australia and who have received support from a hospital-wide transition support service
  Interventions: Behavioral: Transition support service

INTERVENTIONS:
Behavioral: Transition support service — The hospital-wide transition support service provides systematic care coordination for young patients prior to the transfer of care
  Groups: Cohort in Australia

SUMMARY:
At least 12% of children have a chronic disease that requires regular medical follow-up after patients reach legal maturity. This international study aims to provide prospective evidence for improving health and wellbeing outcomes in this population.

The primary hypothesis is that transition readiness will be more strongly associated with adherence to follow-up, fewer emergency visits and continued education than disease severity or chronological age.

The secondary hypothesis is that positive experiences of care will be associated with lower levels of anxiety. Positive care experiences and low anxiety will predict better health-related quality of life during the transition period.

A cohort of 504 young patients will be followed for three years. Patients have been recruited from pediatric hospitals 0-12 months prior to the transfer of care and follow-up will be completed after the patients have been followed for two years in adult healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with a chronic medical condition (duration at least 6 months prior to recruitment)
* Attend care and/or follow-up at either the New Children's Hospital in Helsinki, Finland or the Royal Children's Hospital in Melbourne, Australia in one or more of the following disciplines: endocrinology, gastroenterology, cardiology, rheumatology, neurology, pediatric surgery, nephrology and solid organ transplantation.
* Care to be transferred to adult services within 0-12 months following recruitment

Exclusion Criteria:

* Lack of fluency in study languages (Finnish, Swedish and English)
* Cognitive limitations that inhibit responding to questionnaires

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Researchers approached all eligible patients until 250 patients at both study sites were recruited. According to power calculations, this will be sufficient to have a 90% chance of detecting, as significant at the 5% level, a 5% change in quality of life, even if groups differ in size.
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in 16D health-related quality of life | Baseline to two years post-transfer
  16D is a generic, validated self-report of health related quality of life (HRQoL). It has 16 dimensions, all rated on a 5-point Likert scale. The total 16D score varies from 0 to 1, with 1 being the best imaginable state of HRQoL and with a minimum important change of 0.015.
Change in PedsQL health-related quality of life | Baseline to two years post-transfer
  The Pediatric Quality of Life Inventory (PedsQL) is another validated generic tool to measure HRQoL. It includes 25 questions divided into 4 categories (physical, emotional, social and school). Scores range from 0 to 100, with 100 the best imaginable HRQoL.
Change in health status | Baseline to two years post-transfer
  Patients will report on their symptom severity during the past week using the Visual Analog Scale (VAS). The VAS is a line, 10cm long, with worst imaginable health at one end, and best imaginable health at the other end. Patients make a mark indicating their health between these.
Change in anxiety related to transition of care | Baseline to two years post-transfer
  The State-Trait Anxiety Inventory (STAI) is a validated, 6-item self-report tool to measure anxiety. Items are rated on a 4-point Likert scale. Possible scores range between 20-80, with higher scores indicating higher anxiety.
Missed appointments | Two years post-transfer
  Data linkage will be used to gather the number of missed appointments (uncancelled, not rescheduled) in adult health care. These will serve as one indicator of treatment adherence.
Emergency admissions | Two years post-transfer
  Data linkage will be used to gather information on emergency admissions after the transfer of care. Admissions related to the respective chronic health conditions will serve as one indicator of treatment adherence.

SECONDARY OUTCOMES:
Change in educational status | Baseline to two years post-transfer
  In a questionnaire, patients will annually report on their education status. (Specific question and response options: What is your current education status? Tick one: High school, University student, Homemaker or caregiver, Other (please specify), I'm not enrolled in any studies. These figures will be compared with respective national data.
Change in employment status | Baseline to two years post-transfer
  In a questionnaire, patients will annually report on their employment status. (Specific question and response options: What is your current employment status? Tick one: Working part-time (<30 hours/week); Working full-time (incl. working in shifts); Unemployed, looking for work; Unemployed, not looking for work; Homemaker or caregiver; Other (please specify). These figures will be compared with respective national data.

OTHER OUTCOMES:
Adolescent-friendliness of healthcare services in pediatric and adult hospitals | Baseline to two years post-transfer
  Patients will evaluate the healthcare services they utilize using the Adolescent-friendly hospital survey that was developed in Melbourne in 2011. The survey includes eight items, with four response options each (I fully agree, I somewhat agree, I disagree and I don't know).

CONTACTS AND LOCATIONS:
Locations (2):
- Royal Children's Hospital, Melbourne, Victoria, Australia
- Pediatric Research Center, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
Only collated data may be shared according to EU and Commonwealth data protection requirements.

REFERENCES:
- [Derived] Alanen A, Kallio M, Culnane E, Koivisto M, Pasanen M, Salantera S, Sawyer S, Kosola S. Anxiety and care experiences in adolescents with chronic health conditions: an international, longitudinal study across the transfer of care. BMJ Paediatr Open. 2024 Nov 19;8(1):e002836. doi: 10.1136/bmjpo-2024-002836. PMID 39566994
- [Derived] Kallio MM, Tornivuori A, Kolho KL, Culnane E, Loftus H, Sawyer SM, Kosola S. Changes in health-related quality of life during transition to adult healthcare: an international prospective cohort study. Arch Dis Child. 2024 Jul 18;109(8):659-665. doi: 10.1136/archdischild-2024-327017. PMID 38768988
- [Derived] Kallio M, Tornivuori A, Miettinen PJ, Kolho KL, Relas H, Culnane E, Loftus H, Sawyer SM, Kosola S. Health-related quality of life and self-reported health status in adolescents with chronic health conditions before transfer of care to adult health care: an international cohort study. BMC Pediatr. 2024 Mar 8;24(1):163. doi: 10.1186/s12887-024-04629-x. PMID 38459510
- [Derived] Tornivuori A, Kallio M, Culnane E, Pasanen M, Salantera S, Sawyer S, Kosola S. Transition readiness and anxiety among adolescents with a chronic condition and their parents: A cross-sectional international study. J Adv Nurs. 2024 Feb;80(2):756-764. doi: 10.1111/jan.15860. Epub 2023 Sep 10. PMID 37691321
- [Derived] Kosola S, Culnane E, Loftus H, Tornivuori A, Kallio M, Telfer M, Miettinen PJ, Kolho KL, Aalto K, Raivio T, Sawyer S. Bridge study protocol: an international, observational cohort study on the transition of healthcare for adolescents with chronic conditions. BMJ Open. 2021 Jun 21;11(6):e048340. doi: 10.1136/bmjopen-2020-048340. PMID 34155079